CLINICAL TRIAL: NCT04379830
Title: The Effect of Preoperative Very Low Energy Diet on Mesorectal Volume in Rectal Cancer Patients: A Pilot Study
Brief Title: Preoperative Very Low Energy Diet for Obese Rectal Cancer Patients
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: There were no patients recruited during the trial period. This was a result of: 1) COVID-19 pandemic; 2) MRIs were done prior to patients being seen in consultation, which made them ineligible for enrolment.
Sponsor: McMaster University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 8246
Record Dates: First submitted 2020-04-30; First posted 2020-05-08 (Actual); Last update posted 2024-01-05 (Actual); Status verified 2024-01

CONDITIONS: Rectal Cancer; Obesity
Keywords: Very Low Energy Diet; Low Anterior Resection; Laparoscopy; Magnetic Resonance Imaging
MeSH Terms: conditions — Rectal Neoplasms; Obesity

STUDY DESIGN:
Intervention Model Description: This study is a single center, single-arm prospective cohort pilot study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Very Low Energy Diet (Experimental): VLED in its entirety is composed of the following for 3-weeks preoperatively: Optifast 900 with a single piece of fruit for breakfast, Optifast 900 with one cup of vegetables for lunch, and Optifast 900 with one cup of vegetables for dinner. Patients will be provided written information on fruits and vegetables permitted for consumption with Optifast 900 to provide a total energy intake between 450 and 800 kilocalories (kcal) per day.
  Interventions: Dietary Supplement: Very Low Energy Diet

INTERVENTIONS:
Dietary Supplement: Very Low Energy Diet — Optifast 900 is an FDA approved commercial nutritionally complete meal replacement product manufactured and marketed in the United States. Optifast 900 will be employed as part of the VLED in the present study in the following manner: Optifast 900 with a single piece of fruit for breakfast, Optifast 900 with one cup of vegetables for lunch, and Optifast 900 with one cup of vegetables for dinner. Patients will be provided written information on fruits and vegetables permitted for consumption with Optifast 900 to provide a total energy intake between 450 and 800 kilocalories (kcal) per day.
  Other Names: Optifast 900

SUMMARY:
This pilot study will aim to determine the feasibility, safety, and cost associated with a preoperative VLED for obese rectal cancer patients. Ultimately, the investigators seek to provide evidence that may inform the development of a standardized preoperative weight loss protocol in obese rectal cancer patients.

DETAILED DESCRIPTION:
This study is a single center, single-arm prospective cohort pilot study with a primary aim of determining the feasibility, safety, and cost associated with a preoperative VLED for obese rectal cancer patients. Efficacy of preoperative VLED in this study population will be assessed through measures of mesorectal fat volume with MRI at two separate time points, prior to commencing a pre-operative VLED diet and immediately prior to patients undergoing laparoscopic low anterior resection for rectal cancer, to objectively quantify the proportion of mesorectal fat loss in response to VLED. Secondary aims include an assessment of whether preoperative weight loss contributes to improved intraoperative outcomes including operative time, blood loss, and rate of conversion to open procedure. Furthermore, postoperative outcomes including rates of 30-day complication rate, hospital stay, among others will be evaluated.

Optifast 900 will be administered to enrolled patients over a 3-week period immediately prior to their scheduled elective operation date. Compliance will be measured with a food diary. Two MRIs of the rectum will be obtained: one prior to the commencement of VLED and one following the completion of the VLED before the scheduled operation date. The first MRI will be a clinically indicated preoperative staging investigation, while the second MRI will be used purely for research purposes. Patients will be enrolled in an enhanced recovery after surgery (ERAS) for colorectal surgery program. All patients will be followed by their surgeon as per that individual surgeon's postoperative surveillance schedule. At the routine one-month follow-up visit, patients will see the surgeon as well as a study investigator who will complete a standardized follow up questionnaire, focusing on adverse events and functional independence. Research personnel and study investigators will follow patients throughout their postoperative course in hospital and note any secondary outcomes including laboratory tests or adverse events through the electronic patient chart.

Ultimately, the investigators seek to provide evidence that may inform the development of a standardized preoperative weight loss protocol in obese rectal cancer patients.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* BMI greater than or equal to 30kg/m2 and less than or equal to 55kg/m2
* Patients undergoing elective surgery
* Documented pathological diagnosis of rectal adenocarcinoma
* Preoperative staging investigations consistent with stage I, II, and III disease
* Laparoscopic surgery occurring at St. Joseph's Healthcare Hamilton

Exclusion Criteria:

* BMI less than 30kg/m2
* Contraindications to magnetic resonance imaging, general anesthesia, or major colorectal surgery
* Patient undergoing open surgery
* Patients undergoing emergency or palliative surgery
* Preoperative staging investigations consistent with metastatic disease
* Allergy or contraindication to the use of Optifast
* Prior pelvic colorectal surgery or bariatric surgery
* Enrolled in any other clinical trials or prospective studies where similar outcomes are measured
* Severe, chronic cardiovascular disease (i.e. recent myocardial infarction, unstable angina), renal disease, or hepatic dysfunction
* Patients with pharmacologically managed diabetes mellitus
* Pregnant and/or breastfeeding patients
* Inability to provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-08-01 (Actual); Primary Completion 2023-03-01 (Estimated); Study Completion 2023-06-30 (Estimated)

PRIMARY OUTCOMES:
Recruitment Target (trial feasibility) | 6 months
  20 patients over 6 months (3.33 patients per month)
Medication Compliance Rate (trial feasibility) | 6 months
  Percentage of participants adhering to prescribed Optifast 900 dosages and percentage of Optifast 900 dosages missed by study participants
Follow-Up Rate (trial feasibility) | 6 months
  Percentage of participants completing follow up appointments, questionnaires, and investigations
Incidence of Treatment-Emergent Adverse Events (safety and tolerability) | 2 months
  Change in functional independence from the preoperative, pre-VLED period to 1-month postoperatively using the World Health Organization Disability Assessment Schedule 2.0
Change in Mesorectal Fat Volume (efficacy) | 1 month
  Change in mesolectal fat volume on MRI from prior to 3 weeks of preoperative VLED to immediately following completion of preoperative VLED

SECONDARY OUTCOMES:
Cost | 6 months
  Comparison of the cost (in Canadian dollars) of a 3-week course of Optifast 900 to the cost associated with length of hospital stay and additional treatments during index hospitalization (e.g. reoperation, packed red blood cell transfusion)
Postoperative Length of Stay | 1 month
  Length of stay (LOS) in hospital postoperatively in days
Postoperative Adverse Events | 1 month
  All adverse events attributable to the index surgery for up to 30 days following hospital discharge, including: surgical site infection (SSI), urinary tract infection (UTI), venous thromboembolism (VTE), pneumonia, acute kidney injury (AKI), postoperative ileus, anastomotic leak, wound dehiscence, erectile dysfunction, and readmission
Operative Time | 1 day
  Operative time during index surgery for rectal cancer in minutes
Intraoperative Blood Loss | 1 day
  Blood loss during index surgery for rectal cancer in millilitres
Intraoperative Adverse Events | 1 day
  Review of surgical dictation for any deviation from expected intraoperative processes

CONTACTS AND LOCATIONS:
Locations (1):
- St. Joseph's Healthcare, Hamilton, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No